CLINICAL TRIAL: NCT02797249
Title: Low Dose Aspirin in the Prevention of Preeclampsia in Chinese Pregnant Women.
Brief Title: Low Dose Aspirin in the Prevention of Preeclampsia in China
Acronym: APPEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Li Lin, PhD, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APPEC-2016
Record Dates: First submitted 2016-06-07; First posted 2016-06-13 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Preeclampsia
Keywords: preeclampsia; low dose aspirin; prevention
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspirin (Experimental): Low dose aspirin (100 mg) starting between 12+ and 20 weeks of pregnancy until 34 weeks of pregnancy, taking at night.
  Interventions: Drug: Aspirin
- blank (Other): Routine examination during pregnancy.
  Interventions: Other: Blank

INTERVENTIONS:
Drug: Aspirin — Low dose aspirin（100mg）per day starting between 12+ and 20 weeks of pregnancy until 34 weeks of pregnancy,taking at night.
  Other Names: ASA; acetyl salicylic acid
  Arms: aspirin
Other: Blank — Routine examination during pregnancy.
  Arms: blank

SUMMARY:
Preeclampsia is one of the three leading causes of maternal morbidity and mortality all over the world. The use of low dose aspirin has been mentioned in several studies with promising results. The investigators decided to evaluate the use of low dose aspirin in Chinese pregnant women, starting between 12+ and 20 weeks of pregnancy, based on clinical characteristics aiming to reduce the incidence of preeclampsia.

DETAILED DESCRIPTION:
Detailed Description:

The investigators will conduct a randomized control trial to estimate the efficacy of low dose aspirin in preventing preeclampsia in Chinese pregnant women who are evaluated with risk factors. The investigators will also obtain biological specimen including maternal blood, cord blood, placenta specimen and etc. for basic science studies.

Rationale for Design:There is a lack of evidences or guideline of aspirin using in preventing PE for Chinese women. The investigators will conduct a randomized control trial, which is the 'gold standard' of research design, hoping to answer the question.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age between 12+ and 20 weeks of pregnancy
2. High risk of preeclampsia, based in clinical risk factors as:

   2.1 if they have one or more of the following risk factors： Preeclampsia in a previous pregnancy ,Diabetes Mellitus(Type 1 or 2),Chronic Hypertension .

   2.2 if they have two or more of the following risk factors: Pre-pregnancy Body Mass Index ≥28kg/m2, Elderly pregnancy(age ≥35 years), Mother or sisters with preeclampsia in a previous pregnancy, Primiparity or Famliy history (Mother or sister that developed preeclampsia in a previous pregnancy）.
3. Signed informed consent.

Exclusion Criteria:

1. Allergy to aspirin
2. Asthma
3. Peptic ulcers
4. Severe heart, liver, renal disease who can not burden the experiment
5. Rheumatic immune disease
6. Mental disease
7. Alcohol and drug abuse
8. Being in another drug experiment within 3 months
9. Difficult to follow-up

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Prevention of preeclampsia | 6 months
  The number of cases of preeclampsia that appear in both groups before 34 weeks of pregnancy.

SECONDARY OUTCOMES:
Prevention of preeclampsia at term | 6 months
  The number of cases of preeclampsia that appear in both groups between 37 and 41 weeks of pregnancy.
Fetal Growth Restriction | 6 months
  The number of cases of fetal growth restriction, defined as a fetal weight below the 10th percentile and an abnormal umbilical cord doppler that appear in both groups at any given time during pregnancy.
Preterm birth | 6 months
Abruptio placenta | 6 months
  The number of cases of abruptio placenta that appear in both groups at any given time during pregnancy.
Maternal hemorrhage and neonatal intracranial hemorrhage | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Huixia Yang, PhD, Study Chair — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] LeFevre ML; U.S. Preventive Services Task Force. Low-dose aspirin use for the prevention of morbidity and mortality from preeclampsia: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Dec 2;161(11):819-26. doi: 10.7326/M14-1884. PMID 25200125
- [Background] WHO Recommendations for Prevention and Treatment of Pre-Eclampsia and Eclampsia. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK140561/ PMID 23741776
- [Background] Henderson JT, Whitlock EP, O'Connor E, Senger CA, Thompson JH, Rowland MG. Low-dose aspirin for prevention of morbidity and mortality from preeclampsia: a systematic evidence review for the U.S. Preventive Services Task Force. Ann Intern Med. 2014 May 20;160(10):695-703. doi: 10.7326/M13-2844. PMID 24711050
- [Background] Duley L, Henderson-Smart DJ, Meher S, King JF. Antiplatelet agents for preventing pre-eclampsia and its complications. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004659. doi: 10.1002/14651858.CD004659.pub2. PMID 17443552
- [Background] Visintin C, Mugglestone MA, Almerie MQ, Nherera LM, James D, Walkinshaw S; Guideline Development Group. Management of hypertensive disorders during pregnancy: summary of NICE guidance. BMJ. 2010 Aug 25;341:c2207. doi: 10.1136/bmj.c2207. No abstract available. PMID 20739360
- [Derived] Lin L, Huai J, Li B, Zhu Y, Juan J, Zhang M, Cui S, Zhao X, Ma Y, Zhao Y, Mi Y, Ding H, Chen D, Zhang W, Qi H, Li X, Li G, Chen J, Zhang H, Yu M, Sun X, Yang H. A randomized controlled trial of low-dose aspirin for the prevention of preeclampsia in women at high risk in China. Am J Obstet Gynecol. 2022 Feb;226(2):251.e1-251.e12. doi: 10.1016/j.ajog.2021.08.004. Epub 2021 Aug 10. PMID 34389292
- [Derived] Lin L, Zhu Y, Li B, Yang H; APPEC Study Group. Low-dose aspirin in the prevention of pre-eclampsia in China (APPEC study): protocol for a multicentre randomized controlled trial. Trials. 2018 Nov 6;19(1):608. doi: 10.1186/s13063-018-2970-3. PMID 30400937